CLINICAL TRIAL: NCT02385409
Title: Incidence and Reasons for Preoperative Anemia in Elective Lower Joint Arthroplasty - A Descriptive Study
Brief Title: Incidence and Reasons for Preoperative Anemia in Elective Lower Joint Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Oeivind Jans (Other)
Collaborators: Hvidovre University Hospital (Other)
Responsible Party: Sponsor-Investigator, Oeivind Jans, M.D., Ph.D., Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: RH-4074-OJ5
Record Dates: First submitted 2015-02-16; First posted 2015-03-11 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Anemia; Arthroplasty, Replacement, Hip; Arthroplasty, Replacement, Knee
Keywords: Patient Blood Management; Preoperative anemia; Hip replacement; Knee replacement
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Elective Total Hip- or Knee arthroplasty patients: Patients scheduled for elective Hip- or knee replacement at Hvidovre Hospital, Denmark.

SUMMARY:
Preoperative anemia is an independent risk factor for the need for allogeneic transfusion during surgery and increased postoperative morbidity.

Treatment of preoperative anemia is recommended. However the type of preoperative anemias in elective hip- and knee surgery has only been sparsely studied.

This observational study aims to investigate the incidence and type of anemias prior to elective hip- and knee arthroplasty.

DETAILED DESCRIPTION:
Preoperative anemia is an independent risk factor for the need for allogeneic transfusion during surgery and increased postoperative morbidity.

In elective orthopedic surgery, international guidelines recommends treatment of preoperative anemia including the use of Iron supplements for anemias associated with iron deficiency. In addition, low iron stores in both anemic and non-anemic patients may delay postoperative hemoglobin recovery.

However, the reasons for preoperative anemia and the prevalence of patients with low iron stores have only been sparsely studied in elective hip- and knee arthroplasty.

This observational study aims to investigate the incidence and type of anemias prior to elective hip- and knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Scheduled for elective primary hip- or knee replacement.

Exclusion Criteria:

* Not possible to obtain preoperative blood sample.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients scheduled for elective primary hip- and knee replacement during a 1 year sampling period at the department of orthopedic surgery, Hvidovre Hospital, Denmark
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Anemia Classification - Biochemical classification from preoperative venous blood samples | Date of preoperative blood sampling
  Biochemical classification from preoperative venous blood samples

SECONDARY OUTCOMES:
Prevalence of Anemia according to WHO definitions | Date of preoperative blood sampling
  According to WHO definitions
Proportions of non-anemic patients with low irons stores | Date of preoperative blood sampling
  Low Ferritin or Transferin saturation (TSAT)

CONTACTS AND LOCATIONS:
Overall Officials: Øivind Jans, M.D., Ph.D., Study Director — Rigshospitalet, Denmark
Locations (1):
- Hvidovre Hospital, Department of orthopaedic surgery, Hvidovre, Denmark